CLINICAL TRIAL: NCT03381391
Title: Adapting a Secondary Prevention Program for Nonstudent Emerging Adult Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Cathy Barraco, Associate Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-065; 15-091
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback intervention condition (Experimental)
  Interventions: Behavioral: Personalized Feedback Intervention
- Assessment-only control condition (No Intervention)

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — The current intervention included personalized feedback regarding their alcohol consumption, alcohol-related consequences, gender-specific normative drinking comparisons, personal risk factors (e.g., dependence symptoms, family history of alcoholism), and alcohol expectancies. The intervention also included didactic material related to alcohol (e.g., effects at different BAC levels, tolerance) and drinking moderation strategies. The feedback was presented graphically in a feedback report with the individual's information.
  Arms: Feedback intervention condition

SUMMARY:
Emerging adulthood is a period of heightened vulnerability for problematic alcohol use. Considerable research has been devoted to reducing alcohol risks in college student populations, though far less effort has focused on their noncollege-attending peers. Research targeting nonstudent emerging adults is critical as this group is at risk for experiencing alcohol-related harms. Consequently, the main objective of the present study was to examine the preliminary efficacy of a brief personalized feedback intervention (PFI) tailored for nonstudent at-risk drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Study eligibility included being 18 to 25 years old, having no prior or current college attendance (e.g., technical/vocational programs, associate's degree programs, or four year college programs), and not being currently enrolled in high school. High school completion was not a required eligibility criteria. They also had to report engaging in a minimum of two heavy drinking episodes (i.e., 4/5+ standard drinks for women/men on one occasion) in the past month

Exclusion Criteria:

* Exclusion criteria included consumption above 40 drinks weekly and/or a history of substance use treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 164 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Alcohol use quantity | 9 months
  Alcohol consumption was assessed using the Daily Drinking Questionnaire (DDQ; Collins et al., 1985). Participants reported the number of standard drinks (e.g., 12-ounce beer, 5-ounce wine, or 1.5 ounce liquor) consumed and duration each day during a typical week in the past 3 months. Indices of weekly drinking derived from the DDQ were: total quantity, frequency of drinking days, number of heavy drinking days (days where 4/5+ drinks for women/men were consumed), proportion of heavy drinking days out of total drinking days, maximum number of drinks on the heaviest drinking day, and typical blood alcohol concentration (BAC; see Matthews & Miller, 1979).
Alcohol-related harms | 9 months
  Alcohol-related problems were measured by the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ; Kahler et al., 2005). The B-YAACQ is a 24-item, yes-no format questionnaire assessing negative drinking-related consequences experienced during the past month. Items were summed to create an overall score (ranging from 0 to 24), with higher scores indicating greater severity.